# *Title of the study:*

The effect of personal protective aids on hypertension and diabetes in people exposed to high levels of air pollution

# Date of the document:

January 1, 2021

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

Investigators: Dr. Anubha Goel; Dr. Dweep Barbhaya, Dr. Aditya Khetan, Dr. Jennifer Tran

# **INFORMED CONSENT DOCUMENT**

#### I. Project Title:

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

### II. Introduction/Purpose

You are being asked to participate in this research study because you are part of Dalkhola town where this research study is being conducted. Heart disease is increasingly becoming common in India and the two major risk factors for heart disease are high blood pressure (hypertension) and high blood sugar (diabetes). The purpose of this research study is to study the effects of personal protective aids (air purifier and N95 mask) on blood glucose and blood pressure in communities such as yours.

#### III. Expected Duration of the study and number of research participants:

You will be one of around 150 participants enrolled in this research. Total Duration of study is 10 weeks; however, you will be asked to wear a face mask and use an air purifier for 8 weeks.

#### **IV.** Study Procedures

You will be asked to use an air purifier for 12 hours when you're at home (during the hours of 8 PM to 8 AM) and wear a N-95 mask when you are outdoors (that includes any activity outside your home). You will be given air purifiers and a reusable N95 face mask by our community health workers (CHWs). Our CHWs will train you on how to use them. They will also record your blood glucose and blood pressure every 2 weeks. The study will be divided into 2 parts, 4 weeks each. You'll be in part I for 4 weeks and then will have a break for 2 weeks. Later on, we will put you in part II for 4 weeks; which completes 10 weeks of the study duration. The study will be supervised by local coordinators and investigators.

#### V. Risks and discomforting of patients:

Your participation in this study does not involve any physical risk to you. The puncture of your skin with a lancet to draw blood for measuring your blood sugar can be painful; however, this discomfort is very minimal and brief. For most people, lancet punctures to get blood samples do not cause any serious problems; however, they may cause bleeding, bruising, discomfort, infections, dizziness, or fainting.

#### VI. Benefits

You may not benefit from participation in the study. However, your participation may lead to a better understanding of the benefits of these personal protective devices; which in turn will reduce cardiovascular risk factors (diabetes and hypertension) in the whole community. This might allow doctors to take better care of patients like you. This will also help us provide evidence to policymakers to take strict measure to control air pollution.

#### VII. Financial Information

There is no direct cost to you or your insurance for participation in this study. There will be no financial benefits for participating in the study. CHWs will provide you with air purifiers and N95 face mask. You

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

Investigators: Dr. Anubha Goel; Dr. Dweep Barbhaya, Dr. Aditya Khetan, Dr. Jennifer Tran

will be able to keep the N-95 mask at the end of the study. The indoor air purifier will be collected by the CHW at the end of the study.

#### VIII. Research-Related Injury

There is no risk involved which will lead to research related injury.

#### IX. Summary of your rights as a participant in a research study

Your participation in this research study is voluntary. Refusing to participate will not alter your usual health care or involve any penalty or loss of benefits to which you are otherwise entitled. If you decide to join the study, you may withdraw at any time and for any reason without penalty or loss of benefits. If information generated from this study is published or presented, your identity will not be revealed. In the event new information becomes available that may affect the risks or benefits associated with this study or your willingness to participate in it, you will be notified so that you can decide whether or not to continue participating.

#### X. Confidentiality

All your identifying information such as name, phone number and address will be accessible only to the study personnel (Dweep Barbhaya & Aditya Khetan). This information will be kept safe and confidential by the said personnel. All your data will be stored in a secure database with access only to some of study investigators. The local study investigators will have access to the data, but the data will not be released to government authorities or any person not involved directly with the study. The information will not be revealed unless required by the law.

#### XI. Alternatives to Study Participation

Subjects do not have to participate in the study. Non-participation will not in any way affect you or your relationship with the community and physicians in the community.

#### XII. Disclosure of your study records

Efforts will be made to keep the personal information in your research record private and confidential, but absolute confidentiality cannot be guaranteed. *IIT-Kanpur IRB board may review your study records*. If your records are reviewed, your identity could become known, but only to those authorities concerned with research.

# MIII. Contact information has described to you what is going to be done, the risks, hazards, and benefits involved of participating in the study. The study is being conducted locally by 'Dalkhola SEHAT Welfare Society' and the local site in charge is

The study is being conducted locally by 'Dalkhola SEHAT Welfare Society' and the local site in charge is Dr. Dweep Barbhaya & Dr. Aditya Khetan. They can be contacted at +91-9819403829/+91-9434055047 or by email at <a href="mailto:dweepbarbhaya@gmail.com">dweepbarbhaya@gmail.com</a> or dradityakhetan@gmail.com.

The Principal Investigator, Dr. Anubha Goel, can also be contacted at anubha@iitk.ac.in

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

Investigators: Dr. Anubha Goel; Dr. Dweep Barbhaya, Dr. Aditya Khetan, Dr. Jennifer Tran

If the researchers cannot be reached, or if you would like to talk to someone other than the researcher(s) about concerns regarding the study; research participant's rights; research- related injury; or other human subject issues please contact:

Member Secretary Institution Ethics Committee – IITK, FB - 624, Faculty Building, IIT Kanpur Kanpur - 208016.

#### XIV. Consent:

I have or have had read to me the information given in the informed consent document for this study entitled: "The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution."

- 1. I have received an explanation of the nature, purpose, duration, and foreseeable effects and risks of the trial and what I will be expected to do. My questions have been answered satisfactorily.
- 2. I understand that my participation in the study is voluntary and I may refuse to participate or may withdraw from the trial at any time, without penalty or loss of benefits to which I am otherwise entitled.
- 3. I further understand that any information that becomes available during the course of the study, that may affect my willingness to take part, will be communicated to me.
- 4. Institutional Ethics Authorities may wish to examine my medical records to verify the information collected. By signing this document, I give permission for this review of my records.
- 5. I understand that my identity will not be revealed in any report or publication.
- 6. I agree to take part in above study.

| | <u></u> | | | |
|---|---|---|---|---|
| Name of research participant | Signature/thumb impression of research participants | | nts | Date |
| Name of person Administrating Consent | | Signature of the person administering cons | ent | Date |
| Name of Legal Representative | | Signature of Legal Representative | Dat | te |

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

Investigators: Dr. Anubha Goel; Dr. Dweep Barbhaya, Dr. Aditya Khetan, Supreme Jain

# অবহিত সম্মতি দম্ভাবেজ

# ।. প্রোজেন্ট শিবোনাম:

উদ্দ মাত্রার বায়ু দূষণের সংস্পর্শে আসা লোকদের মধ্যে, উদ্দ রক্তচাপ এবং ডায়াবেটিসের ক্ষেত্রে ব্যক্তিগত প্রতিরক্ষা খুবই প্রভাবকারী।

# **।**।. সুচনা/উদ্দেশ্য

আপনাকে এই গবেষণার সমীক্ষায় অংশ নিতে বলা হচ্ছে কারণ আপনি ডালখোলা শহরে থাকেন যেখানে এই সমীক্ষাটি পরিচালনা করা হচ্ছে। হৃদরোগের সমস্যা ভারতে ক্রমশ সাধারণ হয়ে উঠছে এবং হৃদরোগের জন্য দুটি প্রধান ঝুঁকির কারণ হল উচ্চ রক্ত চাপ/ব্লাড প্রেশার (উচ্চ রক্তচাপ) এবং উচ্চ ব্লাড সুগার (ডায়বেটিক)। এই রিসার্চ সমীক্ষার প্রধান উদ্দেশ্য হল আপনার মতো সম্প্রদায়গুলিতে ব্লাড ফ্লকোজ এবং রক্ত চাপের উপর ব্যক্তিগত সুরক্ষা মূলক সহায়কগুলির (এয়ার পিউরিফায়ার এবং এন 95 মাক্ষ) প্রভাব সম্পর্কে অধ্যয়ন করা।

- াাা. সমীক্ষায় লাগা প্রত্যাশিত সময়কাল এবং গবেষণা অংশগ্রহণকারীদের সংখ্যা: এই সমীক্ষায় আপনি 150 জন তালিকাভুক্ত অংশগ্রহনকারী একজন।এই সমীক্ষায় লাগা সময়কাল হল 10 সপ্তাহ; তবে, আপনাকে ৪ সপ্তাহের জন্য আপনাকে ফেস মাস্ক পড়তে হবে এবং একটি এয়ার পিউরিফায়ার ব্যবহার করতে হবে।
- IV. সমীক্ষার পদ্ধতি

আপনাকে ঘরে থাকাকালীন 12 ঘন্টার (সকাল ৪ টা থেকে রাত ৪ টা অবধি সময় কে ধরা হয়েছে) জন্য এয়ার পিউরিফায়ার ব্যবহার করতে বলা হবে এবং বাইরে বেরোবার(যেটার মধ্যে বাইরে বেরিয়ে করা যেকোনো অ্যাক্টিভিটিকেই ধরা হবে) সময় এন–95 মাস্ক পড়তে বলা হবে।আপনাকে আমাদের সম্প্রদায়ের স্বাস্থ্য কর্মীরা (সিএইচডাবলু)এই এয়ার পিউরিফায়ার এবং পুনরায় ব্যবহারযোগ্য এন–95 মাস্ক দেবেন।আমাদের সম্প্রদায়ের স্বাস্থ্যকর্মীরা (সিএইচডাবলু)এগুলির ব্যবহার কিভাবে করতে হয় সেটা আপনাদের জানিয়ে দেবেন।ভারা আপনার রাড প্লকোজ এবং রাড প্রেশার প্রত্যেক 2 সপ্তাহ অন্তর আসে নিয়ে যাবেন। এই সমীস্কাটি দুটি ভাগে করা হবে, প্রত্যেকটির জন্য 4 সপ্তাহ। আপনি প্রথম ভাগের জন্য 4 সপ্তাহ অংশগ্রহণ করবেন এবং ভারপর আপনাকে 2 সপ্তাহের জন্য ছুটি দেওয়া হবে । ভারপর আবার আপনি দ্বিতীয় ভাগের 4 সপ্তাহের জন্য অংশগ্রহণ করবেন; যেটা শেষ হবে মোট সময়সীমা 10 সপ্তাহে।সমীস্কাটি স্থানীয় সমন্থয়কারী এবং ভদন্তকারীরা দেখাশোনা করবেন।

V. রোগীর ঝুঁকি এবং অসুবিধাঃ

এই সমীক্ষায় আপনার অংশগ্রহনের ফলে আপনার কোন প্রকারের শারীরিক ছ্ষতি হবে না।আপনার রক্তে ফ্লকজের মাত্রা দেখতে ল্যানসেট ফুটিয়ে রক্ত নেওয়ার ক্ষেত্রে হয়তো আপনার একটু কষ্ট হতে পারে; তবে এই কষ্ট খুবই কম এবং স্বল্পছনের জন্য।বেশিরভাগ লোকের ক্ষেত্রে ল্যানসেট ফুটিয়ে রক্ত নেওয়ার ক্ষেত্রে কোন ধরনের কোন গুরুত্তর সমস্যা দেখা দেয় না, তবে এতে রক্তপাত, হ্ষত, অস্বস্থি, সংক্রমণ, মাখা ঘোরা বা অজ্ঞান হয়ে যেতে পারে।

#### VI. উপকারিতা

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

Investigators: Dr. Anubha Goel; Dr. Dweep Barbhaya, Dr. Aditya Khetan, Supreme Jain

আপনি এই সমীক্ষা খেকে হয়তো উপকৃত নাও হতে পারেন। তবে এই সমীক্ষায় আপনার অংশগ্রহণের ফলে এই ব্যক্তিগত সুরক্ষা মূলক ডিভাইসগুলির উপকারিতা সম্পর্কে আরও ভাল ভাবে আমরা বুঝতে পারবো ; যেটার ফলস্বরুপ সমগ্র সম্প্রদায়ের মধ্যে ছদরোগ সংক্রান্ত (মধুমেহ এবং উচ্চরক্তচাপ ) ঝুঁকির সম্ভাবনাগুলি হ্রাস পাবে।এটা চিকিৎসকদের আপনার মতো রোগীদের আরও ভাল ভাবে যত্ন করার অনুমতি দেবে।এটা আমাদের নীতি নির্ধারকদের বায়ু দূষণের পরিমাণ সরবরাহ করতে এবং সেটার নিয়ন্ত্রণে কঠোর ব্যবস্থা নিতে সহায়তা করবে।

# VII. অৰ্থনৈতিক তথ্য

এই সমীক্ষায় আপনার এবং আপনার ইন্সিওরেন্সের সরাসরি কোন মূল্য নেই।এই সমীক্ষায় অংশ নেওয়ার ফলে আপনার কোন প্রকারের কোন আর্থিক সুবিধা হবে না।সিএইচডাবলু রা আপনাকে এয়ার পিউরিফায়ার এবং এন95 ফেস মাস্ক আপনাকে দিয়ে যাবেন।এই সমীক্ষাটির শেষ অবধি আপনি আপনার কাছে এই এন95 ফেস্ক মাস্কটি রাখতে পারবেন।ঘরের জন্য দেওয়া এয়ার পিউরিফায়ারটি সমীক্ষার শেষ অবধি আপনার কাছেই থাকবে যেটা সমীক্ষার শেষে আপনার কাছ থেকে নেওয়া হবে।

VIII. সমীক্ষা সংক্রান্ত ক্ষত এতে কোন প্রকারের কোন ঝুঁকি নেই যেটা সমীক্ষা সম্পর্কিত আঘাতের দিকে পরিচালিত করে।

# IX. সমীক্ষায় একজন অংশগ্রহণকারী হিসাবে আপনার অধিকারের তালিকা

এই সমীক্ষায় আপনার অংশগ্রহণ সম্পূর্ণ আপনার ঐচ্ছিক।এই সমীক্ষায় অংশগ্রহন করতে অশ্বীকার করাতে সেটা কোন ভাবেই আপনার শ্বাভাবিক শ্বাস্থ্য সেবাকে পরিবর্তন করবে না বা কোন ধরণের কোন জরিমানা লাগবে না বা কোন ক্ষতি আপনার হবে না যেটার জন্য আপনি আগে থেকেই যোগ্য।আপনি যদি এই সমীক্ষায় অংশগ্রহণ করবেন বলে সিদ্ধান্ত নেন তাহলে এই সমীক্ষা চলাকালীন যেকোনো সময়ে আপনি এই সমীক্ষাটি প্রত্যাহার করতে পারেন যেকোনো লোকশান বা আপনার প্রাপ্য সুবিধার ক্ষতি ছাড়াই।এই সমীক্ষায় পাওয়া তথ্য উপস্থাপন করার সময় আপনার পরিচয় সম্পূর্ণরূপে গোপন রাখা হবে।এই ইভেন্টে যদি কোন নতুন তথ্য পাওয়া যায় যেটা এই সমীক্ষার সাথে যুক্ত ঝুঁকি বা উপকারিতা বা এটিতে অংশ নেওয়ার আপনার অভিজ্ঞতাকে প্রভাবিত করতে পারে সেক্ষেত্রে আপনাকে জানিয়ে দেওয়া হবে, যাতে আপনি এই সমীক্ষায় অংশগ্রহণ করতে চান কি চান না সেই ব্যাপারে আপনি সিদ্ধান্ত নিতে পারেন।

# X. গোপনীয়তা

আপনার সকল তথ্য যেমন আপনার নাম, ফোন নম্বর এবং ঠিকানা শুধুমাত্র সমীক্ষাকর্মীরাই (দ্বীপ বারভায়া এবং আদিত্য কেতন) দেখতে পারবেন। আপনার সকল প্রকার তথ্য উপরোক্ত কর্মীদের দ্বারা সম্পূর্ণ রূপে গোপন এবং সুরক্ষিত রাখা হবে। স্থানীয় সমীক্ষা তদন্তকারীদের এই ডাটাতে অ্যাক্সেস থাকবে, তবে তথ্যগুলি সরকারি কর্তৃপক্ষের কাছে বা সমীক্ষার সাথে জড়িত কোন ব্যক্তির কাছে প্রকাশ করা হবে না। আইন দ্বারা প্রয়োজনীয় না হলে তথ্য প্রকাশ করা হবে না।

# XI. সমীক্ষায় অংশগ্রহনের বিকল্প

এই সমীক্ষায় বিষয়কে অংশ নিতে হবে না। আপনার অংশগ্রহন না করাটা কোনওভাবেই আপনাকে বা আপনার সম্প্রদায়ের চিকিৎসকদের সাথে আপনার সম্পর্ককে প্রভাবিত করবে না।

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

Investigators: Dr. Anubha Goel; Dr. Dweep Barbhaya, Dr. Aditya Khetan, Supreme Jain

# XII. আপনার সমীষ্ণার রেকর্ড প্রকাশ

সমীক্ষার জন্য করা রেকর্ডে আপনার ব্যক্তিগত তখ্য গোপনীয় রাখার চেষ্টা করা হবে, তবে নিখুঁত ভাবে গোপনীয়তার নিশ্চয়তা দেওয়া যায় না।আইআইটি-কানপুর আইআরবি বোর্ড আপনার সমীক্ষার রেকর্ডটি হয়তো পর্যালোচনা করতে পারে।যদি রেকর্ড পুনরায় দেখা হয় তাহলে আপনার পরিচিতি হয়তো উল্মোচিত হতে পারে, কিক্ত শুধুমাত্র সেই সকল সংস্থার কাছে যারা এই সমীক্ষার সাথে যুক্ত।

#### XIII. যোগাযোগের তথ্য

আপনাকে কী হতে চলেছে , ঝুঁকি, বিপদ এবং সমীক্ষায় অংশ নেওয়ার সাথে জড়িত সুবিধাগুলি কি কি। এই সমীক্ষাটি স্থানীয় ভাবে 'ডালখোলা সেহত কল্যান সমীতি' পরিচালনা করছে এবং স্থানীয় সাইটটির দাযিত্বে আছে ডাকার দ্বীপ বরভ্যা এবং ডাকার আদিত্য খেতান। তাদের সাথে যোগাযোগের নম্বর হল

দায়িত্বে আছে ডাক্তার দ্বীপ বরভয়া এবং ডাক্তার আদিত্য খেতান। তাদের সাথে যোগাযোগের নম্বর হল +91-9819403829/+91-9434055047 বা ইমেল ঠিকানা <u>dweepbarbhaya@gmail.com</u> or <u>dradityakhetan@gmail.com</u> মাধ্যমে যোগাযোগ করা যেতে পারে

প্রিন্সিপাল ইনভেন্টিগেটর ডঃ অনুভা গোয়েলের সাথেও <u>anubha@iitk.ac.in</u>এ যোগাযোগ করা যেতে পারে

যদি সমিক্ষকদের কাছে পৌঁছানো না যায়, বা আপনি সমীক্ষক ব্যাতিত অন্য কারোর সাথে সমীক্ষার সম্পর্কে কথা বলতে ঢান ; সমীক্ষায় অংশগ্রহনকারীদের অধিকার; সমীক্ষা সম্পর্কিত আঘাত;বা অন্যান্য মানব নির্মিত সমস্যা ইত্যাদির সাথে যোগাযোগ করুনঃ

মেম্বার সেক্রেটরি ইন্সটিটিউট এথিক্স কমিটি– আইআইটিকে, এফবি – 624, ফ্যাকাল্টি বিল্ডিং, আইআইটি কানপুর কানপুর – 208016.

## XIV. সম্মতি পত্ৰঃ

এই সমীক্ষার জন্য অবহিত নথিতে দেওয়া সম্মতি তথ্যগুলি আমি পড়েছিঃ
"উদ্ভ রক্তচাপ এবং মধুমেহর ক্ষেত্রে ব্যক্তিগত সুরক্ষামূলক সহায়তার প্রভাব,সেই সকল মানুষদের যারা
অত্যাধিক বায়ু দূষণে থাকেন"।

The effect of personal protective aids on hypertension and diabetes, in people exposed to high levels of air pollution

Investigators: Dr. Anubha Goel; Dr. Dweep Barbhaya, Dr. Aditya Khetan, Supreme Jain

- 1. আমি এই সমীক্ষার প্রকৃতি, উদ্দেশ্য, সময়কাল এবং আগাম প্রভাব এবং ঝুঁকিগুলির ব্যাখ্যা পেয়েছি এবং আমার এটা থেকে কি প্রত্যাশা করা উচিৎ সেটাও জানতে পারেছি। আমার সকল প্রশ্নের সক্তষ্টিজনক উত্তর দেওয়া হয়েছে।
- 2. আমি বুঝতে পেরেছি যে এই সমীক্ষায় আমার অংশগ্রহণ সম্পূর্ণরূপে ঐচ্ছিক এবং আমি অংশ নিতে অস্বীকার করতে পারি বা যেকোনো সময়ে এটার খেকে বেরিয়ে আসতে পারি, কোন পেনাল্টি ছারাই বা আমার প্রাপ্য যেকোন ধরণের সুবিধার ক্ষতি ছাড়াই এটা খেকে সরে আসতে পারি।
- 3. আমি আরও বুঝতে পেরেছি যে সমীক্ষা চলাকালীন এমন কোন তখ্য পাওয়া যায় যেটা যা আমার অংশ করাকে প্রভাবিত করতে পারে,তাহলে আমাকে সেই ব্যাপারে জানানো হবে।
- 4. ইন্সটিটিউশনাল এথিক্স অথরিটিস হয়তো আমার মেডিক্যাল রেকর্ডগুলি পরীক্ষা করে দেখতে পারেন সংগ্রহ করা তথ্য জাচাও করার জন্য।এই ডকিউমেন্টে হস্তাক্ষর করে আমি আমার এই রেকর্ডগুলির পর্যালোচনা করার জন্য অনুমতি দেবো।
- 5. আমি বুঝতে পেরেছি যে কোন রিপোর্ট বা পাব্লিকেশনে আমার পরিচ্য় প্রকাশিত হবে না।
- 6. আমি এই সমীক্ষায় অংশগ্রহণ করতে রাজি।

| সমীক্ষার অংশগ্রহণকারীর নাম | | ——<br>তারিথ |
|---|---|---|
| সম্মতিপত্র পরিচালনাকারী ব্যক্তির নাম | সম্মতিপত্র পরিচালনাকারী ব্যক্তির হস্তাক্ষর | <u> </u> |
| ————————————————————————————————————— | <br>আইনি প্রতিনিধির হস্তাক্ষর | তারিখ |